CLINICAL TRIAL: NCT06491498
Title: Hemidiaphragmatic Paralysis Following Ultrasound-Guided Supraclavicular Brachial Plexus Blockade in Patients Undergoing Upper Limb Surgery
Brief Title: Hemidiaphragmatic Paralysis Following Supraclavicular Brachial Plexus Blockade.
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abanoub Youssief Mosaad, Resident in Anesthesia and ICU department faculty of medicine, Sohag university, Sohag University
Other Study IDs: Soh-Med-24-05-14MS
Record Dates: First submitted 2024-06-03; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Respiratory Depression
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group R in the right upper limb.: Group R (30) will receive 15 mL of 0.5% bupivacaine with dexametomidine by dose 1 μg / kg in the right upper limb.
  Interventions: Diagnostic Test: Supraclavicular Brachial Plexus Blockade
- Groub L in the left upper limb.: Groub L (30) will receive 15 mL of 0.5% bupivacaine with dexametomidine by dose 1 μg / kg in the left upper limb.
  Interventions: Diagnostic Test: Supraclavicular Brachial Plexus Blockade

INTERVENTIONS:
Diagnostic Test: Supraclavicular Brachial Plexus Blockade — Hemidiaphragmatic Paralysis Following Ultrasound-Guided Supraclavicular Brachial Plexus Blockade in patients undergoing upper limb surgery

SUMMARY:
The supraclavicular block is a regional anesthetic technique used as an alternative or adjunct to general anesthesia or used for postoperative pain control for upper extremity surgeries (mid-humerus through the hand). First introduced in 1911 by Kulenkampff as a landmark-based approach, the associated risk of pneumothorax was likely responsible for the technique falling out of favor. With the advent of ultrasonography, La Grange described the utilization of the Doppler probe to identify arteries in 1978. Contemporarily, Kapral and colleagues advocated for the dynamic use of ultrasound to guide needle advancement in the supraclavicular position. Colloquially known as the "spinal of the arm," the supraclavicular block is advantageous as the brachial plexus nerves are tightly packed in this approach and speed of onset is often rapidly achieved. However, because of this consolidated relationship, consider restricting volumes of local anesthesia to as low as possible to achieve goals, as compression ischemia may occur.

DETAILED DESCRIPTION:
The brachial plexus is formed by the anterior primary rami of C5 through T1 and provides sensory and motor innervation of the upper extremity. The brachial plexus is divided, proximally to distally, into rami/roots, trunks, divisions, cords, and terminal branches. The trunks can be found within the posterior triangle of the neck, between the anterior and middle scalene muscles. The brachial plexus, along with the axillary artery, can be considered as a large neurovascular bundle that travels in the axilla to supply the upper extremity.

The brachial plexus provides somatic motor and sensory innervation to the upper extremity, including the scapular region. As the brachial plexus travels through the posterior triangle of the neck into the axilla, arm, forearm, and hand, it contains various named regions based on how the plexus is formed. Ventral rami from spinal nerves C5 through T1, often referred to as roots of the brachial plexus, come together to allow their fibers to intermingle, forming superior, inferior, and middle trunks.

The 3 trunks continue from the posterior triangle into the axilla, with C5 and C6 roots forming the superior trunk, C8 and T1 roots forming the inferior trunk, and the C7 root continuing as the middle trunk.

Continuing from the trunks are bundles that are called divisions. Each of the trunks of the brachial plexus continues as an anterior and posterior division to form lateral, posterior, and medial cords.

The phrenic nerve Comprised of the anterior branches of the C3-C5 spinal roots, the phrenic nerve usually lies on the surface of the anterior scalene muscle underneath the sternocleidomastoid muscle before it enters the thorax behind the subclavian vein, although anatomic variations are common. Because of its close proximity to the brachial plexus, Phrenic nerve palsy (PNP) resulting in ipsilateral hemi diaphragmatic paralysis which can occur following brachial plexus blockade.

Hemi diaphragmatic paralysis (HdP) due to inadvertent phrenic nerve palsy (PNP) is a well-recognized complication of brachial plexus blockade, the incidence of PNP has been reported to be as high as 100% following interscalene brachial plexus block and 50% to 67% following supraclavicular block. While PNP is generally considered rare following infraclavicular block, the incidence prior to the widespread adoption of ultrasound-guided regional anesthesia using solely landmark-based or nerve-stimulator techniques has been reported as high as 26%.

As the brachial plexus and phrenic nerve diverge from each other as they move caudally, ultrasound-guided Supraclavicular Block (SCB) could be a safe, reliable and effective alternative.

Ultrasonography of the diaphragmatic dome is a straight-forward, reliable, non-invasive and reproducible method for assessing the activity of the diaphragm. In fact, Motion- mode can be used to assess diaphragmatic excursion (i.e., displacement) during a voluntary sniff test for which patients forcefully inhaled through the nose in a sniffing fashion. This study will be conducted to evaluate the incidence of hemi diaphragmatic paralysis following ultrasound-guided supraclavicular plexus blockade.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years. American Society of Anesthesiologists physical status 1 to 3, Able to give informed consent. Body mass index (BMI) less than 35.

Exclusion Criteria:

* Patient refusal. Known/suspected allergy to local anesthetics Pregnancy Body mass index (BMI) greater than 35 kg/m2 Neuromuscular disease Obstructive or restrictive pulmonary disease Known or suspected PNP or diaphragmatic dysfunction Other medical or anatomic contraindication to brachial plexus blockade as judged by the investigator

  * local infection.
  * significant coagulation abnormalities.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Age between 18 and 60 years. American Society of Anesthesiologists physical status 1 to 3, Able to give informed consent. Body mass index (BMI) less than 35.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
incidences of hemi diaphragmatic paralysis following ultrasound-guided supraclavicular plexus blockade | 2 hours
  By Using M-mode Ultrasonography showing the limitation of diaphragmatic motion before and after supraclavicular brachial plexus blockade

SECONDARY OUTCOMES:
Evaluation of post operative pain by visual analog scale | 2 hours
  effect on vital signs
Evaluation of oxygen saturation by pulse oximeter | 2 hours
  effect on vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Magdy M Amin, Professor, Principal Investigator — Sohag University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bigeleisen PE. Anatomical variations of the phrenic nerve and its clinical implication for supraclavicular block. Br J Anaesth. 2003 Dec;91(6):916-7. doi: 10.1093/bja/aeg254. PMID 14633767
- [Background] Rose M, Ness TJ. Hypoxia following interscalene block. Reg Anesth Pain Med. 2002 Jan-Feb;27(1):94-6. doi: 10.1053/rapm.2002.29709. PMID 11799511
- [Background] Erickson JM, Louis DS, Naughton NN. Symptomatic phrenic nerve palsy after supraclavicular block in an obese man. Orthopedics. 2009 May;32(5):368. doi: 10.3928/01477447-20090501-02. PMID 19472948
- [Background] Feigl GC, Litz RJ, Marhofer P. Anatomy of the brachial plexus and its implications for daily clinical practice: regional anesthesia is applied anatomy. Reg Anesth Pain Med. 2020 Aug;45(8):620-627. doi: 10.1136/rapm-2020-101435. Epub 2020 May 28. PMID 32471922